CLINICAL TRIAL: NCT03734536
Title: Prospective Multi-center Study Comparing REGENETEN in Lieu of Standard Arthroscopic Repair of High-grade (>50%) Partial-thickness Tears
Brief Title: Treatment of Partial-Thickness Rotator Cuff Tears
Acronym: REGEN PUB 2018
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business reasons not related to patient safety
Sponsor: Smith & Nephew, Inc. (Industry)
Collaborators: Global Research Solutions (Industry); Medical Metrics Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REGEN.PUB.2018.09
Record Dates: First submitted 2018-11-06; First posted 2018-11-08 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2023-10

CONDITIONS: Arthroscopic Surgical Treatment of High-grade (>50%) Partialthickness
Keywords: REGENETEN; REGENETEN Bioinductive Implant; highgrade partial thickness tear; rotator cuff tear; rotator cuff repair
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- REGENETEN™ Bioinductive Implant (Other): Surgical treatment of partial-thickness rotator cuff tears with the REGENETEN Bioinductive Implant system.
  Interventions: Device: REGENETEN™ Bioinductive Implant
- Arthroscopic repair of the high-grade (>50%) partial-thickness (Other): Surgical treatment of partial-thickness rotator cuff tears using standard techniques.
  Interventions: Device: Arthroscopic repair of the high-grade (>50%) partial-thickness

INTERVENTIONS:
Device: REGENETEN™ Bioinductive Implant — The REGENETEN™ Bioinductive Implant is a bioabsorbable device that provides a layer of collagen over injured tendons.
  Arms: REGENETEN™ Bioinductive Implant
Device: Arthroscopic repair of the high-grade (>50%) partial-thickness — Surgical treatment of partial-thickness rotator cuff tears using standard techniques.
  Arms: Arthroscopic repair of the high-grade (>50%) partial-thickness

SUMMARY:
The goal of this clinical trial is to demonstrate that REGENETEN is superior to standard repair techniques when surgically treating high-grade (>50%) partial-thickness tears.

DETAILED DESCRIPTION:
The objective of this study is to demonstrate arthroscopic surgical treatment of high-grade (>50%) partial-thickness tears using REGENETEN yields statistically superior patient post-operative recovery outcomes, faster return to activities of daily living, and less health care utilization versus standard surgical repair techniques.

ELIGIBILITY:
Inclusion Criteria:

Patients will be considered qualified for enrollment if they meet the following criteria:

1. Male or female ≥18 years
2. High-grade (>50% tendon thickness) partial-thickness tear
3. Failed conservative medical management of the tendon tear defined as:

   1. Four (4) to six (6) weeks of formal physical therapy or guided home exercises
   2. Activity modification
   3. Shoulder injection at the discretion of the surgeon
4. Able to comply with the post-operative physiotherapy and follow-up schedule
5. Able to speak and read English Provide written informed consent

Exclusion Criteria:

Any one (1) of the following criteria will disqualify a patient from participation in the study:

1. Prior shoulder surgery on index shoulder within 12 months of enrollment
2. Failed primary rotator cuff surgery of the index shoulder
3. On steroids within 1 month of enrollment
4. Metastatic disease
5. Concomitant surgeries for bone defects requiring bone implantation (Latarjet procedures) or for superior labral tear from anterior to posterior (SLAP)
6. Concomitant biceps tenodesis
7. Rheumatoid arthritis
8. Advanced osteoarthritis
9. Fatty infiltration of the index shoulder rotator cuff muscle ≥ Grade 3
10. Chronic pain disorders (i.e., fibromyalgia)
11. History of insulin dependent diabetes
12. History of heavy smoking (> 1 pack per day) within 6 months of enrollment
13. Currently involved in any injury litigation or workers compensation claims
14. Hypersensitivity to bovine-derived materials Medical or physical condition that, in the opinion of the Investigator, would preclude safe participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Harris, Principal Investigator — Texas Orthopedic Specialists
Locations (10):
- United States (10):
  - University of Florida Orthopaedics and Sports Medicine, Gainesville, Florida
  - Baptist Health, Jacksonville Beach, Florida
  - Harbin Clinic, Rome, Georgia
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Health Center, New Orleans, Louisiana
  - Anne Arundel Medical Center/Luminis Health, Annapolis, Maryland
  - Syracuse Orthopedic Specialist, DeWitt, New York
  - Columbia University, New York, New York
  - Orthopedic Associates of SW Ohio, Centerville, Ohio
  - Texas Orthopedic Specialists, Bedford, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant consented 05 December 2018; study premature termination 14 February 2023 with last participant termination on 11 September 2023.
Pre-assignment Details: There were 168 participants enrolled in the study with 50 participants excluded during surgery or prior to surgery that resulted in 118 participants being treated and allocated into treatment arms.
Period: Overall Study
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Started | 59 | 59
Completed | 48 | 47
Not Completed | 11 | 12
Not completed — Withdrew Consent | 1 | 5
Not completed — Lost to Follow-up | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness | Total
Number analyzed (Participants) | 59 | 59 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.51 (10.57) | 58.98 (8.14) | 55.75 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 33 | 63
  Male | 29 | 26 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race / Ethnicity: White | 55 | 52 | 107
  Race / Ethnicity: Black or African American | 4 | 6 | 10
  Race / Ethnicity: Asian | 0 | 0 | 0
  Race / Ethnicity: American Indian or Alaska Native | 0 | 0 | 0
  Race / Ethnicity: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Race / Ethnicity: African/Caribbean | 0 | 0 | 0
  Race / Ethnicity: Other | 0 | 0 | 0
  Race / Ethnicity: Missing | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 59 | 59 | 118
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.08 (8.30) | 29.41 (4.81) | 30.25 (6.80)
Index shoulder [Count of Participants; unit: Participants]
  Left | 19 | 28 | 47
  Right | 40 | 31 | 71
  Not Reported | 0 | 0 | 0
Prescription opioid or non-opioid pain medication use to manage pain other than index shoulder pain [Count of Participants; unit: Participants] — Previous treatment that occurred pre-index shoulder surgery (i.e., before the surgical treatment identified for this study)
  Participants
    No | 0 | 0 | 0
    Yes | 6 | 5 | 11
    Missing | 53 | 54 | 107
Surgery on Dominant Arm [Count of Participants; unit: Participants]
  Yes | 22 | 24 | 46
  No | 12 | 25 | 37
  Missing | 25 | 10 | 35
Treatment to Manage Index Shoulder: Prescription Non-Opioid Pain Medication [Count of Participants; unit: Participants] — Previous treatment that occurred pre-index shoulder surgery (i.e., before the surgical treatment identified for this study)
  Participants
    No | 44 | 40 | 84
    Yes | 15 | 19 | 34
    Missing | 0 | 0 | 0
Treatment to Manage Index Shoulder: Prescription Opioid Pain Medication [Count of Participants; unit: Participants] — Previous treatment that occurred pre-index shoulder surgery (i.e., before the surgical treatment identified for this study)
  Participants
    No | 56 | 51 | 107
    Yes | 3 | 8 | 11
    Missing | 0 | 0 | 0
Treatment to Manage Index Shoulder: Steroid Injection(s) [Count of Participants; unit: Participants] — Previous treatment that occurred pre-index shoulder surgery (i.e., before the surgical treatment identified for this study)
  Participants
    No | 29 | 28 | 57
    Yes | 30 | 31 | 61
    Missing | 0 | 0 | 0
Treatment to Manage Index Shoulder: Shoulder Surgery [Count of Participants; unit: Participants] — Previous treatment that occurred pre-index shoulder surgery (i.e., before the surgical treatment identified for this study)
  Participants
    No | 55 | 57 | 112
    Yes | 4 | 2 | 6
    Missing | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: American Shoulder and Elbow Surgeons (ASES) Score
Description: American Shoulder and Elbow Surgeons (ASES) score at baseline and 3 months following index surgery. ASES is composed of 2 sections containing participant self-reported and clinician assessments. The ASES score is a 0 to 100-point rating based solely on participant responses and is a combination of the participant's shoulder pain rating (VAS Pain) and self-reported ability to perform 10 different activities of daily living (ADLs). A higher score is a better outcome.
Time Frame: Baseline and 3 months
Population: Overall number of participants with available data for each treatment at the time frame indicated
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 58 | 56
score on a scale
  Baseline: number analyzed (Participants) | 55 | 56
  Baseline | 59.46 (17.07) | 52.10 (15.61)
  3 months | 80.07 (13.30) | 74.61 (12.35)

2. Secondary Outcome: American Shoulder and Elbow Surgeons (ASES) Score Weekly Through 3 Months Post-Index Surgery
Description: American Shoulder and Elbow Surgeons (ASES) score at baseline and every week up to 12 weeks (3 months) post-index surgery. ASES is composed of 2 sections containing participant self-reported and clinician assessments. The ASES score is a 0 to 100-point rating based solely on participant responses and is a combination of the participant's shoulder pain rating (VAS Pain) and self-reported ability to perform 10 different activities of daily living (ADLs). A higher score is a better outcome.
Time Frame: Baseline, Week 1, Week 2,Week 3,Week 4,Week 5,Week 6,Week 7,Week 8,Week 9,Week 10,Week 11, & Week 12
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 58 | 56
score on a scale
  Baseline: number analyzed (Participants) | 55 | 56
  Baseline | 59.46 (17.07) | 52.10 (15.61)
  Week 1: number analyzed (Participants) | 54 | 53
  Week 1 | 49.00 (13.42) | 44.42 (11.22)
  Week 2: number analyzed (Participants) | 57 | 55
  Week 2 | 54.77 (13.04) | 50.04 (12.92)
  Week 3: number analyzed (Participants) | 57 | 55
  Week 3 | 57.67 (13.65) | 51.77 (12.62)
  Week 4: number analyzed (Participants) | 58 | 54
  Week 4 | 60.22 (12.69) | 51.77 (11.19)
  Week 5: number analyzed (Participants) | 55 | 53
  Week 5 | 63.90 (12.91) | 56.89 (9.84)
  Week 6: number analyzed (Participants) | 56 | 55
  Week 6 | 66.25 (13.05) | 59.06 (11.77)
  Week 7: number analyzed (Participants) | 57 | 54
  Week 7 | 66.72 (14.42) | 62.18 (12.66)
  Week 8: number analyzed (Participants) | 57 | 53
  Week 8 | 70.74 (13.98) | 63.74 (11.98)
  Week 9: number analyzed (Participants) | 55 | 55
  Week 9 | 73.70 (13.94) | 66.05 (12.54)
  Week 10: number analyzed (Participants) | 55 | 56
  Week 10 | 76.81 (11.43) | 69.62 (11.69)
  Week 11: number analyzed (Participants) | 57 | 53
  Week 11 | 78.14 (11.94) | 71.80 (13.43)
  Week 12 | 80.07 (13.30) | 74.61 (12.35)

3. Secondary Outcome: Single Assessment Numeric Value (SANE) Score Weekly Through 3 Months Post-Index Surgery
Description: Single Assessment Numeric Evaluation (SANE) score at baseline and weekly up to 12 weeks (3 months). SANE scores range from 0 to 100, with 100 indicating a better outcome. SANE is a simple, patient-based shoulder function assessment tool measured by answering a single question:
  ''How would you rate your shoulder today as a percentage of normal (0% to 100% scale with 100% being normal)?''
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11, Week 12
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 59 | 59
score on a scale
  Baseline | 47.42 (21.34) | 36.78 (17.90)
  Week 1: number analyzed (Participants) | 55 | 53
  Week 1 | 28.22 (21.63) | 17.85 (17.23)
  Week 2: number analyzed (Participants) | 57 | 55
  Week 2 | 35.37 (20.93) | 24.27 (17.86)
  Week 3: number analyzed (Participants) | 57 | 53
  Week 3 | 39.89 (18.79) | 31.94 (16.35)
  Week 4: number analyzed (Participants) | 59 | 55
  Week 4 | 45.73 (16.76) | 42.27 (17.18)
  Week 5: number analyzed (Participants) | 55 | 54
  Week 5 | 49.00 (17.18) | 40.19 (18.56)
  Week 6: number analyzed (Participants) | 58 | 55
  Week 6 | 54.60 (16.83) | 42.27 (17.18)
  Week 7: number analyzed (Participants) | 57 | 55
  Week 7 | 56.35 (18.59) | 46.56 (16.48)
  Week 8: number analyzed (Participants) | 57 | 53
  Week 8 | 59.91 (19.88) | 49.77 (15.81)
  Week 9: number analyzed (Participants) | 55 | 55
  Week 9 | 61.82 (18.22) | 53.55 (15.17)
  Week 10: number analyzed (Participants) | 56 | 55
  Week 10 | 67.66 (16.23) | 57.27 (15.15)
  Week 11: number analyzed (Participants) | 57 | 53
  Week 11 | 69.86 (14.80) | 59.45 (18.04)
  Week 12: number analyzed (Participants) | 58 | 56
  Week 12 | 73.31 (16.38) | 63.89 (16.11)

4. Secondary Outcome: American Shoulder and Elbow Surgeons Visual Analog Scale (ASES-VAS) Pain Score Weekly Through 3 Months Post-Index Surgery
Description: Participant reported shoulder pain was measured using the American Shoulder and Elbow Surgeons Visual Analog Scale (AES-VAS) Pain score at baseline and every week up to 12 weeks (3 months) post-index surgery. ASES-VAS Pain scores range from 0 to 10, where 0 indicates no pain and 10 indicates the worst possible pain (i.e., a lower score is a better outcome).
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11, Week 12
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 58 | 56
score on a scale
  Baseline: number analyzed (Participants) | 55 | 56
  Baseline | 4.35 (2.54) | 5.49 (2.49)
  Week 1: number analyzed (Participants) | 54 | 53
  Week 1 | 3.53 (2.27) | 4.15 (2.23)
  Week 2: number analyzed (Participants) | 58 | 55
  Week 2 | 3.03 (2.14) | 3.49 (2.02)
  Week 3: number analyzed (Participants) | 58 | 55
  Week 3 | 2.65 (2.10) | 3.29 (2.25)
  Week 4: number analyzed (Participants) | 58 | 54
  Week 4 | 2.42 (2.09) | 3.34 (1.98)
  Week 5: number analyzed (Participants) | 58 | 53
  Week 5 | 2.32 (1.99) | 2.84 (1.64)
  Week 6: number analyzed (Participants) | 58 | 55
  Week 6 | 2.15 (1.94) | 2.77 (1.90)
  Week 7: number analyzed (Participants) | 58 | 54
  Week 7 | 2.20 (2.13) | 2.58 (1.90)
  Week 8: number analyzed (Participants) | 58 | 53
  Week 8 | 1.79 (2.01) | 2.41 (1.66)
  Week 9: number analyzed (Participants) | 58 | 55
  Week 9 | 1.57 (1.91) | 2.41 (1.73)
  Week 10 | 1.32 (1.55) | 1.97 (1.58)
  Week 11: number analyzed (Participants) | 58 | 53
  Week 11 | 1.27 (1.62) | 1.92 (2.00)
  Week 12 | 1.31 (1.83) | 1.79 (1.75)

5. Secondary Outcome: American Shoulder and Elbow Surgeons (ASES) Score at Baseline, 6 Months, 12 Months, 18 Months and 24 Months
Description: American Shoulder and Elbow Surgeons (ASES) score at baseline, 6, 12, 18 and 24 months following index surgery. ASES is composed of 2 sections containing participant self-reported and clinician assessments. The ASES score is a 0 to 100-point rating based solely on participant responses and is a combination of the participant's shoulder pain rating (VAS Pain) and self-reported ability to perform 10 different activities of daily living (ADLs). A higher score is a better outcome.
Time Frame: Baseline, 6 months, 12 months, 18 months and 24 months
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 55 | 56
score on a scale
  Baseline | 59.46 (17.07) | 52.10 (15.61)
  6 months: number analyzed (Participants) | 55 | 52
  6 months | 90.38 (11.73) | 87.42 (11.25)
  12 months: number analyzed (Participants) | 47 | 49
  12 months | 90.83 (16.55) | 91.98 (12.90)
  18 months: number analyzed (Participants) | 50 | 39
  18 months | 94.71 (13.07) | 92.87 (13.40)
  24 months: number analyzed (Participants) | 47 | 25
  24 months | 94.77 (13.76) | 94.17 (11.76)

6. Secondary Outcome: Single Assessment Numeric Value (SANE) Score at Baseline, 6 Months, 12 Months, 18 Months and 24 Months
Description: Single Assessment Numeric Evaluation (SANE) score at baseline, 6, 12, 18 and 24 months following index surgery. SANE scores range from 0 to 100, with 100 indicating a better outcome. SANE is a simple, patient-based shoulder function assessment tool measured by answering a single question:
  ''How would you rate your shoulder today as a percentage of normal (0% to 100% scale with 100% being normal)?''
Time Frame: Baseline, 6 months, 12 months, 18 months and 24 months
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 59 | 59
score on a scale
  Baseline | 47.42 (21.34) | 36.78 (17.90)
  6 months: number analyzed (Participants) | 51 | 52
  6 months | 86.18 (12.47) | 81.15 (14.12)
  12 months: number analyzed (Participants) | 48 | 49
  12 months | 87.27 (17.35) | 87.86 (14.64)
  18 months: number analyzed (Participants) | 50 | 39
  18 months | 91.74 (12.52) | 90.03 (10.30)
  24 months: number analyzed (Participants) | 48 | 25
  24 months | 90.67 (19.17) | 94.20 (8.07)

7. Secondary Outcome: American Shoulder and Elbow Surgeons Visual Analog Scale (ASES-VAS) Pain Score at Baseline, 6 Months, 12 Months, 18 Months and 24 Months
Description: Participant reported shoulder pain was measured using the American Shoulder and Elbow Surgeons Visual Analog Scale (AES-VAS) Pain score at baseline, 6, 12, 18 and 24 months following index surgery. ASES-VAS Pain scores range from 0 to 10, where 0 indicates no pain and 10 indicates the worst possible pain (i.e., a lower score is a better outcome).
Time Frame: Baseline, 6 months, 12 months, 18 months and 24 months
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 55 | 56
score on a scale
  Baseline | 4.35 (2.54) | 5.49 (2.49)
  6 months: number analyzed (Participants) | 51 | 52
  6 months | 0.79 (1.56) | 0.89 (1.38)
  12 months: number analyzed (Participants) | 47 | 49
  12 months | 1.09 (2.12) | 0.68 (1.62)
  18 months: number analyzed (Participants) | 50 | 39
  18 months | 0.50 (1.56) | 0.77 (1.75)
  24 months: number analyzed (Participants) | 47 | 25
  24 months | 0.48 (1.61) | 0.47 (1.15)

8. Secondary Outcome: Constant-Murley Score at Baseline, 3 Months, 6 Months, 12 Months, and 24 Months
Description: Constant-Murley Score at baseline, 3, 6, 12, and 24 months following index surgery. The Constant-Murley Score is a validated assessment of pain and shoulder functionality. The test is divided into four subscales: pain, activities of daily living, strength, and range of motion (forward elevation, external rotation, abduction, and internal rotation of the shoulder). Constant-Murley Scores range from 0 to 100, with higher scores indicating better shoulder function & lower scores indicating worse shoulder function.
Time Frame: Baseline, 3 months, 6 months, 12 months, and 24 months
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 48 | 50
score on a scale
  Baseline: number analyzed (Participants) | 30 | 50
  Baseline | 53.73 (15.81) | 45.40 (14.13)
  3 months: number analyzed (Participants) | 33 | 43
  3 months | 60.73 (12.05) | 52.35 (12.08)
  6 months: number analyzed (Participants) | 42 | 45
  6 months | 66.10 (10.57) | 61.13 (11.62)
  12 months: number analyzed (Participants) | 48 | 46
  12 months | 69.33 (11.11) | 66.24 (12.45)
  24 months: number analyzed (Participants) | 46 | 22
  24 months | 71.76 (8.65) | 71.18 (9.08)

9. Secondary Outcome: Weekly Opioid Use to Treat Index Shoulder Through 3 Months Post-Index Surgery
Description: Opioid prescription medication use to treat the index shoulder post-index surgery was measured directly after surgery and weekly for up to 12 weeks (3 months) as the total number of defined daily doses (DDD). Participants recorded their use of opioid pain medication in a log within their diary. The total number of DDD was calculated by multiplying the total quantity of the drug (e.g., number of tablets) by the strength (e.g., milligrams per tablet) to obtain the total dosage (e.g., total number of milligrams), then dividing by the World Health Organization (WHO) specified defined daily dose.
Time Frame: Directly after surgery, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11, Week 12
Population: Overall number of participants with available data for the treatment and time frame indicated. One extreme outlier was excluded from the Arthroscopic repair treatment group due to a data irregularity. Only medications with an assigned WHO-specified daily dose were included in the analysis, as the calculation of the total number of defined daily doses (DDD) depends on this value. Medications without a WHO-assigned daily dose value were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: defined daily dose
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 22 | 27
defined daily dose
  Directly after surgery | 7.82 (22.93) | 3.10 (7.53)
  Week 1: number analyzed (Participants) | 17 | 27
  Week 1 | 18.28 (42.90) | 4.22 (10.93)
  Week 2: number analyzed (Participants) | 17 | 19
  Week 2 | 4.38 (6.12) | 1.73 (2.05)
  Week 3: number analyzed (Participants) | 6 | 18
  Week 3 | 3.85 (3.21) | 3.35 (5.12)
  Week 4: number analyzed (Participants) | 6 | 13
  Week 4 | 2.81 (1.64) | 2.58 (2.20)
  Week 5: number analyzed (Participants) | 3 | 11
  Week 5 | 1.17 (0.85) | 1.97 (2.01)
  Week 6: number analyzed (Participants) | 2 | 8
  Week 6 | 0.97 (0.99) | 1.98 (2.04)
  Week 7: number analyzed (Participants) | 0 | 7
  Week 7 |  | 1.56 (2.44)
  Week 8: number analyzed (Participants) | 0 | 1
  Week 8 |  | 0.66 (NA) — Standard Deviation could not be calculated due to insufficient participant data available
  Week 9: number analyzed (Participants) | 0 | 3
  Week 9 |  | 2.11 (1.71)
  Week 10: number analyzed (Participants) | 0 | 1
  Week 10 |  | 2.50 (NA) — Standard Deviation could not be calculated due to insufficient participant data available
  Week 11: number analyzed (Participants) | 0 | 2
  Week 11 |  | 2.34 (2.35)
  Week 12: number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Weekly Non-Opioid Use to Treat Index Shoulder Through 3 Months Post-Index Surgery
Description: Non-opioid prescription medication use to treat the index shoulder post-index surgery was measured directly after surgery and weekly for up to 12 weeks (3 months) as the total number of defined daily doses (DDD). Participants recorded their use of non-opioid pain medication in a log within their diary. The total number of DDD was calculated by multiplying the total quantity of the drug (e.g., number of tablets) by the strength (e.g., milligrams per tablet) to obtain the total dosage (e.g., total number of milligrams), then dividing by the World Health Organization (WHO) specified defined daily dose.
Time Frame: as for outcome 9
Population: Overall number of participants with available data for the treatment and time frame indicated. Only medications with an assigned WHO-specified daily dose were included in the analysis, as the calculation of the total number of defined daily doses (DDD) depends on this value. Medications without a WHO-assigned daily dose value were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: defined daily dose
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 7 | 11
defined daily dose
  Directly after surgery: number analyzed (Participants) | 7 | 8
  Directly after surgery | 6.94 (3.20) | 2.67 (0.89)
  Week 1: number analyzed (Participants) | 4 | 11
  Week 1 | 10.50 (7.67) | 4.21 (6.24)
  Week 2: number analyzed (Participants) | 6 | 5
  Week 2 | 10.50 (8.71) | 5.05 (6.86)
  Week 3: number analyzed (Participants) | 2 | 5
  Week 3 | 20.00 (0) | 3.47 (2.79)
  Week 4: number analyzed (Participants) | 2 | 9
  Week 4 | 20.00 (0) | 1.48 (0.87)
  Week 5: number analyzed (Participants) | 3 | 11
  Week 5 | 14.78 (9.05) | 4.22 (3.85)
  Week 6: number analyzed (Participants) | 3 | 8
  Week 6 | 13.83 (10.68) | 5.63 (3.96)
  Week 7: number analyzed (Participants) | 3 | 8
  Week 7 | 14.00 (10.39) | 5.17 (3.48)
  Week 8: number analyzed (Participants) | 3 | 2
  Week 8 | 15.83 (7.22) | 6.75 (7.42)
  Week 9: number analyzed (Participants) | 3 | 4
  Week 9 | 16.00 (4.00) | 5.01 (5.20)
  Week 10: number analyzed (Participants) | 2 | 3
  Week 10 | 12.00 (11.31) | 5.83 (4.86)
  Week 11: number analyzed (Participants) | 1 | 2
  Week 11 | 20.00 (NA) — Standard Deviation could not be calculated due to insufficient participant data available | 5.17 (5.42)
  Week 12: number analyzed (Participants) | 1 | 2
  Week 12 | 27.00 (NA) — Standard Deviation could not be calculated due to insufficient participant data available | 11.27 (15.18)

11. Secondary Outcome: Opioid Use to Treat the Index Shoulder Directly After Surgery, 6 Months, and 12 Months
Description: Opioid prescription medication use to treat the index shoulder post-index surgery was measured directly after surgery, 6 months, and 12 months as the total number of defined daily doses (DDD). Participants recorded their use of opioid pain medication in a log within their diary. The total number of DDD was calculated by multiplying the total quantity of the drug (e.g., number of tablets) by the strength (e.g., milligrams per tablet) to obtain the total dosage (e.g., total number of milligrams), then dividing by the World Health Organization (WHO) specified defined daily dose.
Time Frame: Directly after surgery, 6 months, and 12 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: defined daily dose
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 22 | 27
defined daily dose
  Directly after surgery | 7.82 (22.93) | 3.10 (7.53)
  6 months: number analyzed (Participants) | 1 | 0
  6 months | 2.40 (NA) — Standard Deviation could not be calculated due to insufficient participant data available |
  12 months: number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Non-Opioid Prescription Medication Use to Treat the Index Shoulder Directly After Surgery, 6 Months, and 12 Months
Description: Non-opioid prescription medication use to treat the index shoulder post-index surgery was measured directly after surgery, 6 months, and 12 months as the total number of defined daily doses (DDD). Participants recorded their use of non-opioid pain medication in a log within their diary. The total number of DDD was calculated by multiplying the total quantity of the drug (e.g., number of tablets) by the strength (e.g., milligrams per tablet) to obtain the total dosage (e.g., total number of milligrams), then dividing by the World Health Organization (WHO) specified defined daily dose.
Time Frame: Directly after surgery, 6 months, and 12 months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: defined daily dose
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 7 | 11
defined daily dose
  Directly after surgery | 6.94 (3.20) | 2.67 (0.89)
  6 months: number analyzed (Participants) | 1 | 1
  6 months | 3.20 (NA) — Standard Deviation could not be calculated due to insufficient participant data available | 19.00 (NA) — Standard Deviation could not be calculated due to insufficient participant data available
  12 months: number analyzed (Participants) | 0 | 1
  12 months |  | 2.00 (NA) — Standard Deviation could not be calculated due to insufficient participant data available

13. Secondary Outcome: Duration of Shoulder Immobilization
Description: Duration of shoulder immobilization measured as days spent in a sling
Time Frame: Following index surgery, up to 7 weeks
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 53 | 50
days | 18.40 (14.55) | 35.72 (12.55)

14. Secondary Outcome: Number of Participants Return to Work Status by Type of Work at 12 Months Post-Index Surgery
Description: Participants ability to return to previous type of work within 12 months post-index surgery was measured by the number of participants work status. Work status was identified as "Not currently employed", "Did not return to work", "Returned to partial, modified, or parttime employment", or "Returned to fulltime employment." The type of work for each work status (excluding "Not currently employed") was then categorized as:
  * Very heavy work
  * Heavy work
  * Medium work
  * Light work
  * Sedentary work
Time Frame: Up to 12 months
Population: Overall number of participants with available data for the treatment and time frame indicated. It was possible for participants to return to partial, modified, or part-time employment, and then return to fulltime employment within the 12 month period. Meaning, multiple responses were allowed.
Measure: Count of Participants; unit: Participants
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 48 | 49
Participants
  Not currently employed | 16 | 20
  Did not return to work : Very heavy work | 0 | 0
  Did not return to work : Heavy work | 0 | 0
  Did not return to work : Medium work | 0 | 1
  Did not return to work : Light work | 0 | 0
  Did not return to work : Sedentary work | 0 | 0
  Returned to partial, modified, or parttime employment : Very heavy work | 0 | 0
  Returned to partial, modified, or parttime employment : Heavy work | 5 | 2
  Returned to partial, modified, or parttime employment : Medium work | 6 | 4
  Returned to partial, modified, or parttime employment : Light work | 3 | 3
  Returned to partial, modified, or parttime employment : Sedentary work | 2 | 3
  Returned to fulltime employment : Very heavy work | 2 | 0
  Returned to fulltime employment : Heavy work | 4 | 5
  Returned to fulltime employment : Medium work | 8 | 7
  Returned to fulltime employment : Light work | 10 | 7
  Returned to fulltime employment : Sedentary work | 8 | 11

15. Secondary Outcome: Time to Return to Driving
Description: Time to return to driving post-index surgery measured in days.
Time Frame: Following index surgery, up to 139 days
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 53 | 48
days | 18.3 (21.60) | 24.54 (19.85)

16. Secondary Outcome: Time to Return to Sports
Description: Time to return to sports involving overhead throwing post-index surgery measured in days.
Time Frame: Following index surgery, approximately 1 year
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 8 | 2
days | 202 (87.18) | 93.50 (17.68)

17. Secondary Outcome: Number of Participants With Progression to Full-Thickness Tear at 12 Months
Description: The number of participants with progression to full-thickness tear at 24 months post-index surgery were identified by supraspinatus imagining of the tear location. The rotator cuff tear was classified as bursal (Yes/No), then categorized as one of the following:
  * Tendinosis
  * Low-grade Partial Thickness Tear
  * High-grade Partial Thickness Tear
  * Full-Thickness Tear
  * Intact
Time Frame: 12 months
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 49 | 48
Participants
  Bursal=Yes | Tendinosis | 7 | 8
  Bursal=Yes | Low-grade Partial Thickness Tear | 6 | 5
  Bursal=Yes | High-grade Partial Thickness Tear | 7 | 5
  Bursal=Yes | Full-Thickness Tear | 1 | 2
  Bursal=Yes | Intact | 2 | 1
  Bursal=No | Tendinosis | 5 | 7
  Bursal=No | Low-grade Partial Thickness Tear | 12 | 6
  Bursal=No | High-grade Partial Thickness Tear | 6 | 5
  Bursal=No | Full-Thickness Tear | 0 | 0
  Bursal=No | Intact | 3 | 9

18. Secondary Outcome: Number of Participants With Progression to Full-Thickness Tear at 24 Months
Description: as for outcome 17
Time Frame: 24 months
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 47 | 21
Participants
  Bursal=Yes | Tendinosis | 10 | 4
  Bursal=Yes | Low-grade Partial Thickness Tear | 5 | 2
  Bursal=Yes | High-grade Partial Thickness Tear | 3 | 2
  Bursal=Yes | Full-Thickness Tear | 1 | 0
  Bursal=Yes | Intact | 3 | 0
  Bursal=No | Tendinosis | 5 | 4
  Bursal=No | Low-grade Partial Thickness Tear | 13 | 6
  Bursal=No | High-grade Partial Thickness Tear | 3 | 1
  Bursal=No | Full-Thickness Tear | 0 | 0
  Bursal=No | Intact | 4 | 2

19. Secondary Outcome: Number of Participants Percent Filling of Rotator Cuff at 12 Months
Description: The number of participants percent filling of the rotator cuff was identified by supraspinatus imagining of the tear location at 12 months post-index surgery as bursal (Yes/No), then categorized as one of the following:
  * 0% to < 25%
  * 25% to < 50%
  * 50% to < 75%
  * 75% to <100%
  * 100%
Time Frame: 12 months
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 33 | 41
Participants
  Bursal=Yes | 0% to < 25% | 1 | 3
  Bursal=Yes | 25% to < 50% | 1 | 0
  Bursal=Yes | 50% to < 75% | 2 | 1
  Bursal=Yes | 75% to < 100% | 6 | 7
  Bursal=Yes | 100% | 4 | 4
  Bursal=No | 0% to < 25% | 1 | 4
  Bursal=No | 25% to < 50% | 5 | 2
  Bursal=No | 50% to < 75% | 2 | 3
  Bursal=No | 75% to < 100% | 10 | 6
  Bursal=No | 100% | 1 | 11

20. Secondary Outcome: Number of Participants Percent Filling of Rotator Cuff at 24 Months
Description: The number of participants percent filling of the rotator cuff was identified by supraspinatus imagining of the tear location at 24 months post-index surgery as bursal (Yes/No), then categorized as one of the following:
  * 0% to < 25%
  * 25% to < 50%
  * 50% to < 75%
  * 75% to <100%
  * 100%
Time Frame: 24 months
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 33 | 20
Participants
  Bursal=Yes | 0% to < 25% | 0 | 3
  Bursal=Yes | 25% to < 50% | 0 | 0
  Bursal=Yes | 50% to < 75% | 0 | 1
  Bursal=Yes | 75% to < 100% | 6 | 3
  Bursal=Yes | 100% | 7 | 1
  Bursal=No | 0% to < 25% | 2 | 0
  Bursal=No | 25% to < 50% | 3 | 1
  Bursal=No | 50% to < 75% | 3 | 1
  Bursal=No | 75% to < 100% | 10 | 5
  Bursal=No | 100% | 2 | 5

21. Secondary Outcome: Rotator Cuff Tendon Thickness at 12 Months
Description: Rotator cuff tendon thickness in millimeters (mm) at 12 months post-index surgery categorized as:
  * Total Thickness (where tendon thickness cannot be differentiated)
  * Thickness of Native (where tendon thickness can be differentiated)
  * Thickness of New Tissue (where tendon thickness can be differentiated)
  * Total Thickness (where tendon thickness can be differentiated)
Time Frame: 12 Months
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 47 | 47
millimeters (mm)
  Total Thickness (where tendon thickness cannot be differentiated): number analyzed (Participants) | 43 | 40
  Total Thickness (where tendon thickness cannot be differentiated) | 4.45 (1.86) | 4.57 (1.75)
  Thickness of Native (where tendon thickness can be differentiated): number analyzed (Participants) | 4 | 7
  Thickness of Native (where tendon thickness can be differentiated) | 3.50 (0.85) | 1.87 (1.13)
  Thickness of New Tissue (where tendon thickness can be differentiated): number analyzed (Participants) | 4 | 7
  Thickness of New Tissue (where tendon thickness can be differentiated) | 2.40 (0.42) | 2.53 (0.79)
  Total Thickness (where tendon thickness can be differentiated): number analyzed (Participants) | 4 | 7
  Total Thickness (where tendon thickness can be differentiated) | 5.90 (0.77) | 4.40 (1.60)

22. Secondary Outcome: Rotator Cuff Tendon Thickness at 24 Months
Description: Rotator cuff tendon thickness in millimeters (mm) at 24 months post-index surgery categorized as:
  * Total Thickness (where tendon thickness cannot be differentiated)
  * Thickness of Native (where tendon thickness can be differentiated)
  * Thickness of New Tissue (where tendon thickness can be differentiated)
  * Total Thickness (where tendon thickness can be differentiated)
Time Frame: 24 Months
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 46 | 21
millimeters (mm)
  Total Thickness (where tendon thickness cannot be differentiated): number analyzed (Participants) | 42 | 19
  Total Thickness (where tendon thickness cannot be differentiated) | 4.88 (1.90) | 4.63 (1.47)
  Thickness of Native (where tendon thickness can be differentiated): number analyzed (Participants) | 4 | 2
  Thickness of Native (where tendon thickness can be differentiated) | 4.00 (0.91) | 2.80 (1.13)
  Thickness of New Tissue (where tendon thickness can be differentiated): number analyzed (Participants) | 4 | 2
  Thickness of New Tissue (where tendon thickness can be differentiated) | 2.38 (0.41) | 2.90 (0.85)
  Total Thickness (where tendon thickness can be differentiated): number analyzed (Participants) | 4 | 2
  Total Thickness (where tendon thickness can be differentiated) | 6.38 (0.90) | 5.70 (0.28)

23. Secondary Outcome: Number of Participants Goutallier Classification of Rotator Cuff at 12 Months
Description: The Goutallier classification was used to classify the fatty infiltration of the rotator cuff. The Goutallier classification ranges from a grade of 0 indicating a completely normal muscles without any fatty streaks to a grade of 4 which indicates that more fat than muscle is present. The number of participants Goutallier classification grade of the rotator cuff at 12 months post-index surgery were identified by supraspinatus imagining of the tear location. The rotator cuff tear was identified as bursal (Yes/No), then classified as one of the following:
  * Grade 1
  * Grade 2
  * Grade 3
  * Grade 4
  * Grade 0
Time Frame: 12 months
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 49 | 48
Participants
  Bursal=Yes | Grade 1 | 15 | 13
  Bursal=Yes | Grade 2 | 1 | 2
  Bursal=Yes | Grade 3 | 0 | 0
  Bursal=Yes | Grade 4 | 0 | 0
  Bursal=Yes | Grade 0 | 7 | 6
  Bursal=No | Grade 1 | 12 | 16
  Bursal=No | Grade 2 | 3 | 4
  Bursal=No | Grade 3 | 0 | 0
  Bursal=No | Grade 4 | 0 | 0
  Bursal=No | Grade 0 | 11 | 7

24. Secondary Outcome: Number of Participants Goutallier Classification of Rotator Cuff at 24 Months
Description: The Goutallier classification was used to classify the fatty infiltration of the rotator cuff. The Goutallier classification ranges from a grade of 0 indicating a completely normal muscles without any fatty streaks to a grade of 4 which indicates that more fat than muscle is present. The number of participants Goutallier classification grade of the rotator cuff at 24 months post-index surgery were identified by supraspinatus imagining of the tear location. The rotator cuff tear was identified as bursal (Yes/No), then classified as one of the following:
  * Grade 1
  * Grade 2
  * Grade 3
  * Grade 4
  * Grade 0
Time Frame: 24 months
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 47 | 21
Participants
  Bursal=Yes | Grade 1 | 13 | 6
  Bursal=Yes | Grade 2 | 1 | 0
  Bursal=Yes | Grade 3 | 0 | 0
  Bursal=Yes | Grade 4 | 0 | 0
  Bursal=Yes | Grade 0 | 8 | 2
  Bursal=No | Grade 1 | 11 | 7
  Bursal=No | Grade 2 | 3 | 3
  Bursal=No | Grade 3 | 0 | 0
  Bursal=No | Grade 4 | 0 | 0
  Bursal=No | Grade 0 | 11 | 3

25. Secondary Outcome: Number of Participants Sugaya Score of Rotator Cuff at 12 Months
Description: The Sugaya score was used to measure the rotator cuff integrity. The Sugaya score ranges from Type I to Type V. Type I indicates a repaired cuff that had sufficient thickness with homogeneously low intensity on the MRI image while Type V indicates the presence of a major discontinuity on the MRI images suggesting a medium or large tear. The number of participants Sugaya Score of the rotator cuff at 12 months post-index surgery were identified by supraspinatus imagining of the tear location. The rotator cuff tear was identified as bursal (Yes/No), then classified as one of the following:
  * Type I
  * Type II
  * Type III
  * Type IV
  * Type V
Time Frame: 12 months
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 47 | 47
Participants
  Bursal=Yes | Type I | 4 | 4
  Bursal=Yes | Type II | 8 | 8
  Bursal=Yes | Type III | 8 | 6
  Bursal=Yes | Type IV | 1 | 2
  Bursal=Yes | Type V | 0 | 0
  Bursal=No | Type I | 6 | 11
  Bursal=No | Type II | 12 | 10
  Bursal=No | Type III | 8 | 6
  Bursal=No | Type IV | 0 | 0
  Bursal=No | Type V | 0 | 0

26. Secondary Outcome: Number of Participants Sugaya Score of Rotator Cuff at 24 Months
Description: The Sugaya score was used to measure the rotator cuff integrity. The Sugaya score ranges from Type I to Type V. Type I indicates a repaired cuff that had sufficient thickness with homogeneously low intensity on the MRI image while Type V indicates the presence of a major discontinuity on the MRI images suggesting a medium or large tear. The number of participants Sugaya Score of the rotator cuff at 24 months post-index surgery were identified by supraspinatus imagining of the tear location. The rotator cuff tear was identified as bursal (Yes/No), then classified as one of the following:
  * Type I
  * Type II
  * Type III
  * Type IV
  * Type V
Time Frame: 24 months
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 45 | 21
Participants
  Bursal=Yes | Type I | 5 | 1
  Bursal=Yes | Type II | 10 | 5
  Bursal=Yes | Type III | 4 | 2
  Bursal=Yes | Type IV | 1 | 0
  Bursal=Yes | Type V | 0 | 0
  Bursal=No | Type I | 7 | 3
  Bursal=No | Type II | 14 | 8
  Bursal=No | Type III | 4 | 2
  Bursal=No | Type IV | 0 | 0
  Bursal=No | Type V | 0 | 0

27. Secondary Outcome: Number of Participants With Revision Surgery
Description: Incidence of revision surgery measured by the number of participants with Revision Surgery (Yes/No) defined as any revision surgery involving the index shoulder for any cause within 24 months post-index surgery.
Time Frame: Following index surgery, up to 24 months
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 59 | 59
Participants
  Revision Surgery: Yes | 1 | 4
  Revision Surgery: No | 58 | 55

28. Secondary Outcome: Aggregate Health Care Utilization Costs
Description: Related health care utilization costs over 12 months post- surgery will be calculated based on health care utilization as reported in the participant diary and/or in the participant's medical records.
Time Frame: Following index surgery, up to 12 months
Population: Appropriate data not collected to perform analysis as a result of study termination
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Operating Room Time (Index Surgery)
Description: Operating time for the index surgery, defined as the time from first incision to wound closure (measured in minutes) as recorded in the operative procedure notes.
Time Frame: Intra-operative
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 55 | 59
minutes | 46.89 (19.13) | 57.05 (19.16)

30. Secondary Outcome: Number of Steroid Injections
Description: The number of steroid injections per participant administered to the index shoulder over 12 months post-index surgery as reported in the participant diary and/or in the participant's medical record.
Time Frame: Following index surgery, up to 12 months
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Mean (Standard Deviation); unit: injections
Units Other Than Participants: injections
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 12 | 10
Number analyzed (injections) | 19 | 16
injections | 1.58 (1.00) | 1.60 (1.00)

31. Secondary Outcome: Number of Unscheduled Clinic Visits
Description: The number of unscheduled clinic visits per participant (defined as a return visit to a health care provider for examination/evaluation of the index shoulder) over 12 months post-index surgery, as reported in the participant diary and/or in the participant's medical record.
Time Frame: Following index surgery, up to 12 months
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Mean (Standard Deviation); unit: unscheduled visits
Units Other Than Participants: unscheduled visits
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 52 | 45
Number analyzed (unscheduled visits) | 214 | 232
unscheduled visits | 4.1 (1.94) | 5.16 (2.08)

32. Secondary Outcome: Number of For-Cause Imaging Procedures
Description: The total number of for cause imaging procedures (e.g., MRI or ultrasound) per participant performed on the index shoulder over 12 months post-index surgery, as reported in the participant diary and/or in the participant's medical record
Time Frame: Following index surgery, up to 12 months
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Mean (Standard Deviation); unit: for-cause imaging procedures
Units Other Than Participants: for-cause imaging procedures
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 11 | 10
Number analyzed (for-cause imaging procedures) | 25 | 15
for-cause imaging procedures | 2.27 (2.28) | 1.50 (0.85)

33. Secondary Outcome: Number of Physiotherapy Sessions
Description: The total number of physiotherapy sessions per participant over 12 months post-index surgery, as reported in the participant diary and/or in the participant's medical record
Time Frame: Following index surgery, up to 12 months
Population: Overall number of participants with available data for the treatment and time frame indicated.
Measure: Mean (Standard Deviation); unit: physiotherapy sessions
Units Other Than Participants: physiotherapy sessions
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
Number analyzed (Participants) | 42 | 45
Number analyzed (physiotherapy sessions) | 773 | 1253
physiotherapy sessions | 18.40 (8.23) | 27.84 (13.41)

ADVERSE EVENTS:
Time Frame: Adverse events were collected upon implantation of device through study termination, up to 2 years
Arm/Group | REGENETEN™ Bioinductive Implant | Arthroscopic Repair of the High-grade (>50%) Partial-thickness
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 33/59 | 17/59
Other Adverse Events (participants affected / at risk) | 51/59 | 56/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | REGENETEN™ Bioinductive Implant (N=59) | Arthroscopic Repair of the High-grade (>50%) Partial-thickness (N=59)
Acute Myeloid Leukemia in Relapse (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute Pyelonephritis (Renal and urinary disorders) | 0 | 1
acute respiratory failure and covid-19 pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
acute respiratory failure, pneumonia, and left pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Adhesive capsulitis left shoulder (Musculoskeletal and connective tissue disorders) | 0 | 1
atherosclerotic occlusive coronary artery disease (Cardiac disorders) | 1 | 0
Avascular Necrosis {left shoulder, hip, ankle with concomitant medial malleolar stress fracture} (Musculoskeletal and connective tissue disorders) | 1 | 0
Candidal Skin Infection (Infections and infestations) | 1 | 0
Cellulitis of Right Upper Extremity (Infections and infestations) | 1 | 0
Chemotherapy Induced Nausea (General disorders) | 1 | 0
COVID-19 (Hospitalization) (Infections and infestations) | 0 | 1
Covid-19, Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cytomegalovirus (Infections and infestations) | 1 | 0
Deep Vein Thrombosis and Superficial Venous Thrombosis of Left Upper Extremity (Vascular disorders) | 0 | 1
epigastric pain with vomiting; anal fistula (Gastrointestinal disorders) | 1 | 0
Failure of Left total knee replacement, subsequent encounter (Musculoskeletal and connective tissue disorders) | 0 | 1
Failure of RIGHT total knee replacement, subsequent encounter (Musculoskeletal and connective tissue disorders) | 0 | 1
Graft vs Host Disease (Immune system disorders) | 1 | 0
infection of left elbow (Infections and infestations) | 1 | 0
Labial Lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Left Knee internal derangement of posterior horn medial meniscus (Musculoskeletal and connective tissue disorders) | 1 | 0
Left knee tibial plateau fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
left lower extremity cellulitis status post coronary artery bypass (Infections and infestations) | 1 | 0
left shoulder arthrofibrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
left shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Left shoulder partial rotator cuff tear (non-study arm) (Injury, poisoning and procedural complications) | 1 | 0
Left Side Pulmonary Embolism (Cardiac disorders) | 1 | 0
Multiple Pulmonary Nodules/Lesions (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neutropenic Fever (Immune system disorders) | 1 | 0
Noninsulin Dependent Diabetes Mellitus with Hyperglycemia (Endocrine disorders) | 1 | 0
Non-ST Elevation Myocardial Infarction (Cardiac disorders) | 0 | 1
Pancytopenia due to Chemotherapy (Blood and lymphatic system disorders) | 1 | 0
Planned Hospital admission for FLU/CY/TBI Haplo AllSCT for AML (Infections and infestations) | 1 | 0
Planned Hospital admit for Cycle 1 of HiDose APA-c (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Postprocedural Bulbous Urethral Stricture (Renal and urinary disorders) | 1 | 0
Pulmonary Embolism (Vascular disorders) | 1 | 0
revision repair of ventral incisional hernia (Gastrointestinal disorders) | 0 | 1
Right Anterior supraspinatus recurrent supraspinatus tear status post prior repair (Musculoskeletal and connective tissue disorders) | 0 | 1
Right carpal tunnel syndrome and right trigger thumb (Musculoskeletal and connective tissue disorders) | 1 | 0
right deltoid muscle strain progressed to rotator cuff re-tear (Musculoskeletal and connective tissue disorders) | 0 | 1
Right inguinal hernia (Gastrointestinal disorders) | 0 | 1
Right Knee Anteromedial Osteoarthritis (Blood and lymphatic system disorders) | 0 | 1
right rotator cuff repair revision with bicep repair (Musculoskeletal and connective tissue disorders) | 0 | 1
Right Rotator cuff tear (Musculoskeletal and connective tissue disorders) | 1 | 0
Right Shoulder Pain Status post Fall (Injury, poisoning and procedural complications) | 1 | 0
Severe iron deficiency anemia requiring blood transfusion (Metabolism and nutrition disorders) | 1 | 0
Unknown dental issue requiring tooth extraction (Surgical and medical procedures) | 0 | 1
unstable angina (Vascular disorders) | 1 | 0
Ureteral Calculus (Renal and urinary disorders) | 1 | 0
Urinary Tract Infection (Renal and urinary disorders) | 2 | 0
ventral hernia (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | REGENETEN™ Bioinductive Implant (N=59) | Arthroscopic Repair of the High-grade (>50%) Partial-thickness (N=59)
Abscess of Right Axilla (Infections and infestations) | 1 | 0
Acute Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Allergic Reaction of unknown origin -Likely food related (Immune system disorders) | 0 | 1
alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Ankle sprain (Injury, poisoning and procedural complications) | 0 | 1
Back muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bilateral biceps tendinitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bilateral Headaches (Nervous system disorders) | 1 | 0
Bilateral Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Blurry Vision (Eye disorders) | 1 | 0
Bronchitis and sinus infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
chronic regional pain syndrome (Nervous system disorders) | 0 | 1
chronic right shoulder pain status post fall, possible adhesive capsulitis (Injury, poisoning and procedural complications) | 1 | 0
Clostridioides Difficile Diarrhea (Infections and infestations) | 1 | 0
Colonoscopy to determine cause of increased diarrhea and stomach pain (Surgical and medical procedures) | 1 | 0
contact dermatitis from surgical tape (Injury, poisoning and procedural complications) | 1 | 0
cough, diarrhea, muscle pain, weakness (General disorders) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 4
decrease range of motion right shoulder (Musculoskeletal and connective tissue disorders) | 1 | 0
dermatitis from surgical bandages (Injury, poisoning and procedural complications) | 0 | 1
Dizziness (Ear and labyrinth disorders) | 1 | 0
Due to dehydration, patient fell. She had mild soreness in index shoulder. (Injury, poisoning and procedural complications) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Elevated liver enzymes - fatty liver (Hepatobiliary disorders) | 0 | 1
Food poisoning/stomach infection/inflamed intestines (Gastrointestinal disorders) | 0 | 1
Fractured Rib after Fall (Injury, poisoning and procedural complications) | 0 | 1
Gout Flare up to Left Ankle (Musculoskeletal and connective tissue disorders) | 1 | 0
Gross Hematuria (Renal and urinary disorders) | 1 | 0
hematuria (Renal and urinary disorders) | 1 | 0
Herpes Simplex Virus Infection ( Right Upper Lip) (Infections and infestations) | 1 | 0
Hypokalemia (Blood and lymphatic system disorders) | 1 | 0
Hypophosphatemia (Blood and lymphatic system disorders) | 1 | 0
Increased left bicep and shoulder pain after increased PT/"bursitis" type symptoms (Musculoskeletal and connective tissue disorders) | 0 | 1
Increased left shoulder pain after fall into wall (Injury, poisoning and procedural complications) | 0 | 1
Increased left shoulder pain after overuse (Injury, poisoning and procedural complications) | 0 | 1
Increased left shoulder pain after slipping in shower and grabbing bar with left arm. (Injury, poisoning and procedural complications) | 0 | 1
Increased left shoulder pain, especially when lifting arm out to the side (Musculoskeletal and connective tissue disorders) | 0 | 1
Increased left shoulder stiffness and pain (Musculoskeletal and connective tissue disorders) | 0 | 1
left AC Joint pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Left Adhesive Capsulitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Left foot arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Left mild tendinopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
left rotator cuff tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Left shoulder biceps tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Left shoulder bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Left shoulder impingement (Musculoskeletal and connective tissue disorders) | 0 | 1
left shoulder osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
left shoulder pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Left shoulder pain after napping without sling (Injury, poisoning and procedural complications) | 0 | 1
left shoulder pain from fall (Injury, poisoning and procedural complications) | 1 | 4
left shoulder pain secondary to a partial thickness bursal sided rotator cuff retear (Injury, poisoning and procedural complications) | 1 | 0
Left shoulder soreness/pain when raising arm to mid-chest level (Musculoskeletal and connective tissue disorders) | 0 | 1
Left wrist pain with numbness in fingers. Carpal tunnel-like symptoms. (Musculoskeletal and connective tissue disorders) | 0 | 1
lumbar pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Lyme disease (Infections and infestations) | 0 | 1
Mucositis due to Antineoplastic Therapy (Injury, poisoning and procedural complications) | 1 | 0
Muscle cramps in left shoulder (Musculoskeletal and connective tissue disorders) | 0 | 1
Myofascial pain around left mid-scapular border (Musculoskeletal and connective tissue disorders) | 0 | 1
new onset pain and motion loss left shoulder due to over-exerting left shoulder (Injury, poisoning and procedural complications) | 1 | 0
Pain under right arm, in armpit area (Musculoskeletal and connective tissue disorders) | 0 | 1
Patient Fall (Injury, poisoning and procedural complications) | 0 | 1
Patient felt a pop and acute increased pain in right shoulder (Injury, poisoning and procedural complications) | 1 | 0
Peripheral Neuropathy (Nervous system disorders) | 1 | 0
primary headache syndrome (Nervous system disorders) | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0
Pseudomonas Urinary Tract Infection (Renal and urinary disorders) | 1 | 0
Rash in Adult located on Left Scapula area (Skin and subcutaneous tissue disorders) | 1 | 0
Respiratory Syncytial Virus (Infections and infestations) | 1 | 0
right acromioclavicular Joint arthritris (Musculoskeletal and connective tissue disorders) | 1 | 0
Right Adhesive Capsulitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Right biceps tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Right Flank Pain (Renal and urinary disorders) | 1 | 0
Right great toe stress fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Right hand gamekeeper's thumb (Musculoskeletal and connective tissue disorders) | 0 | 1
right hip bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
right knee osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Right partial thickness rotator cuff tear (Musculoskeletal and connective tissue disorders) | 1 | 0
right shoulder AC Joint osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Right Shoulder Adhesive Capsulitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Right Shoulder Adhesive Capsulitis/ anterior shoulder pain (impingement) (Musculoskeletal and connective tissue disorders) | 0 | 1
Right shoulder impingement syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
right shoulder pain (Musculoskeletal and connective tissue disorders) | 4 | 2
right shoulder pain due to flare up of biceps tenotomy (Musculoskeletal and connective tissue disorders) | 1 | 0
right shoulder pain from fall (Injury, poisoning and procedural complications) | 1 | 1
Right shoulder pain from physical therapy (Musculoskeletal and connective tissue disorders) | 0 | 1
right shoulder stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Right shoulder tendinosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Right thumb trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0
Right Upper Extremity Hematoma (Skin and subcutaneous tissue disorders) | 1 | 0
Sciatica down right leg (Nervous system disorders) | 0 | 1
Sinus Infection (Infections and infestations) | 0 | 1
Skin lesion on right foot 4th toe (Skin and subcutaneous tissue disorders) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Tremors of right upper extremity (Nervous system disorders) | 1 | 0
Unspecified Lump in the Left Breast (Reproductive system and breast disorders) | 1 | 0
Vaginitis (Reproductive system and breast disorders) | 0 | 1
Vasovagal episode/fall causing broken nose (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Yeast infection (Infections and infestations) | 0 | 1

LIMITATIONS AND CAVEATS:
1. Study terminated due to patient selection bias (age, tear severity).
2. Low patient diary completion compliance (pain medication, for-cause imaging).
3. Unreliable MRI data (ex: tendon fill-in, tendon differentiation, tendon thickness) provided by independent reviewer.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right to modify any proposed publication within 30 days after receipt if it discloses potentially patentable items, patent, trade secret, or other proprietary or confidential information of Sponsor. If patentable items are involved, proposed, disclosure to third party may be delayed up to 90 days. If not submitted within 18 months after the Study's conclusion, the Site/Investigator may publish results after Sponsor's review.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT03734536/Prot_SAP_000.pdf